CLINICAL TRIAL: NCT04703491
Title: A Novel and Adaptive Software for Automated Delivery of Cognitive Behavioral Therapy
Brief Title: TreadWill, an Automated Intervention for Depressive Symptoms
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Indian Institute of Technology Kanpur (Other)
Responsible Party: Principal Investigator, Nitin Gupta, Associate Professor, Indian Institute of Technology Kanpur
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: IITK/IEC/2019-20/II/4
Record Dates: First submitted 2020-12-30; First posted 2021-01-11 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-05

CONDITIONS: Depressive Symptoms
Keywords: depression; anxiety; CCBT; CBM; chatbot; CBT; mindfulness
MeSH Terms: conditions — Depression; Anxiety Disorders | interventions — Drug Interactions

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The participant is masked to the intervention assigned to them. All outcome measures are self-reported by the participants through a computer program without any involvement of the experimenters.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Full intervention (Experimental): This group receives the full-featured intervention, including CCBT, CBM, Mindfulness, chatbot with many interactive elements.
  Interventions: Behavioral: Interactive and full-featured intervention
- Limited CCBT control group (Active Comparator): This group receives feature-limited intervention (text-based computerized CBT)
  Interventions: Behavioral: Feature-limited CCBT
- Waitlist control group (Other): This group receives waitlist control.
  Interventions: Other: Waitlist control

INTERVENTIONS:
Behavioral: Interactive and full-featured intervention — Participants will go through an automated program. Participants will learn and practice the techniques of CBT through multimedia elements. They will play games based on Cognitive Bias Modification (CBM) paradigms, practice mindfulness, and chat with an automated empathic chatbot.
  Arms: Full intervention
Behavioral: Feature-limited CCBT — Participants will be going through an automated program. Participants will learn and practice the techniques of CBT in a plain-text format with reduced features
  Arms: Limited CCBT control group
Other: Waitlist control — Participants will be put on a waitlist for a period of 6 weeks.
  Arms: Waitlist control group

SUMMARY:
TreadWill is a fully automated digital intervention that provides a multi-modal treatment for depressive symptoms. It includes:

1. Slides and interactive text-based conversations based on Cognitive Behavioral Therapy (CBT);
2. Mindfulness videos;
3. Game-based Cognitive Bias Modification paradigms;
4. An empathetic chatbot. This study's primary aim is to test the differential effectiveness of this full-featured version of TreadWill compared to a text-based CBT program.

DETAILED DESCRIPTION:
TreadWill is an online tool to deliver automated intervention for depressive symptoms. TreadWill helps the participants learn the concepts of Cognitive Behavioral Therapy (CBT), and practice mindfulness in an interactive manner. It also has games based on Cognitive Bias Modification (CBM) and an empathetic chatbot. We hypothesize that participants using TreadWill will show a significant reduction in depressive symptoms and will show engagement with the program. To test this hypothesis, we are conducting a randomized controlled trial. We will randomize participants into three groups: experimental, active control, and waitlist. Participants randomized to the experimental group will get access to the full-featured version of TreadWill as described above. Participants randomized to the active control group will have access to a limited version of TreadWill designed to deliver basic CBT in plain text format. The waitlisted participants will be put on a waitlist for 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Fluent in English
* PHQ-9 Score from 5 to 19
* Access to an internet-enabled Android smartphone
* Plan to use TreadWill in Google Chrome browser
* Agree to allow notifications from TreadWill
* Agree to add TreadWill to Home screen
* Have email on one of the HTML-enabled platforms including Gmail, Outlook, Yahoo, Rediffmail, AOL, Hotmail.

Exclusion Criteria:

* Suicide ideation (score greater than 0 on the 9th question of PHQ-9 and score greater than 4 on SIQ)
* Unemployed
* Current or previous diagnosis of bipolar disorder/manic-depressive disorder or psychosis
* Prospective participants who say they only want to check out the program and do not plan to complete it are excluded.
* Used an earlier version of TreadWill

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 500 (Estimated)
Dates: Start 2021-04-27 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Change in Patient Health Questionnaire-9 score | change from baseline to program completion or last usage (upto 90 days).
  Standard questionnaire for depressive symptoms. Total score is used; lower score indicates better outcome.

SECONDARY OUTCOMES:
Change in Generalized Anxiety Disorder 7 score | baseline, post-completion or last usage (upto 90 days), 90 day follow-up after completion
  Standard questionnaire for generalized anxiety symptoms. Total score is used; lower score indicates better outcome.
Time spent with the program | from beginning till study completion date (expected within 1 year from the trial start date)
  Automated measure of time spent on the program for experimental and active comparator group
Follow-up Patient Health Questionnaire-9 score | 90-120 days after program completion
  Standard questionnaire for depressive symptoms. Total score is used; lower score indicates better outcome.

OTHER OUTCOMES:
Change in Patient Health Questionnaire-9 score (Intermediate reports) | after modules 1 (average 1 week), 2 (average 2 weeks), 3 (average 3 weeks), 4 (average 4 weeks) and 5 (average 5 weeks)
  Standard questionnaire for depressive symptoms. Total score is used; lower score indicates better outcome.
Change in Generalized Anxiety Disorder 7 score (Intermediate reports) | after modules 1 (average 1 week), 2 (average 2 weeks), 3 (average 3 weeks), 4 (average 4 weeks) and 5 (average 5 weeks)
  Standard questionnaire for generalized anxiety symptoms. Total score is used; lower score indicates better outcome.
User experience survey | after module 3 (average 3 weeks) and module 6 (upto 90 days) of program
  Computerized survey to get user feedback on the features of the program.
Time spent in playing games | from beginning till study completion date (expected within 1 year from the trial start date)
  Measurement of the total time for which games are played (in seconds).
Frequency of playing games | from beginning till study completion date (expected within 1 year from the trial start date)
  The total number of times for which the games were played
Feedback on the games | from beginning till study completion date (expected within 1 year from the trial start date)
  The number of upvotes and downvotes received on games.
Change in mood during the program | from beginning till study completion date (expected within 1 year from the trial start date)
  Users in the experimental group, using the chatbot, will indicate their mood in one of the three categories: positive, neutral, and negative.
Change in completion of worksheets | from beginning till study completion date (expected within 1 year from the trial start date)
  Automated measure of number of worksheets completed for experimental and active comparator group.
Use of personalization in the chatbot | from beginning till study completion date (expected within 1 year from the trial start date)
  The number of times the users change their preferred frequencies of modules in the chatbot.

CONTACTS AND LOCATIONS:
Overall Officials: Nitin Gupta, PhD, Principal Investigator — Indian Institute of Technology Kanpur
Locations (1):
- Indian Institute of Technology Kanpur, Kanpur, Uttar Pradesh, India

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gilbody S, Brabyn S, Lovell K, Kessler D, Devlin T, Smith L, Araya R, Barkham M, Bower P, Cooper C, Knowles S, Littlewood E, Richards DA, Tallon D, White D, Worthy G; REEACT collaborative. Telephone-supported computerised cognitive-behavioural therapy: REEACT-2 large-scale pragmatic randomised controlled trial. Br J Psychiatry. 2017 May;210(5):362-367. doi: 10.1192/bjp.bp.116.192435. Epub 2017 Mar 2. PMID 28254959
- [Background] Andrews G, Basu A, Cuijpers P, Craske MG, McEvoy P, English CL, Newby JM. Computer therapy for the anxiety and depression disorders is effective, acceptable and practical health care: An updated meta-analysis. J Anxiety Disord. 2018 Apr;55:70-78. doi: 10.1016/j.janxdis.2018.01.001. Epub 2018 Feb 1. PMID 29422409
- See also: Link for TreadWill study — https://www.treadwill.org/iitk